CLINICAL TRIAL: NCT03947190
Title: Safety, Immunogenicity, and Efficacy of R21/Matrix-M and ChAd63/MVA-ME-TRAP in the Context of Controlled Human Malaria Infection: A Phase IIb Trial in Kenyan Adults
Brief Title: A Study to Determine if New Types of Malaria Vaccines Are Safe, Effective and Lead to Immunity in Kenyan Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to US FDA hold on the challenge agent and funding concerns
Sponsor: University of Oxford (Other)
Collaborators: Kenya Medical Research Institute (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC074
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2022-09

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Injections, Intradermal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1 adults (n=24) will be receiving, 4 weeks apart, three doses of 10µg R21 /50µg Matrix M vaccine, and a CHMI intradermally (ID) by inoculation of 22,500 PfSPZ Challenge.
  Interventions: Biological: R21/Matrix-M; Biological: intradermal injection (ID) or direct venous injection (DVI) of PfSPZ Challenge
- Group 2 (Experimental): Group 2 adults (n=24) will be receiving 5x10^10 vp ChAd63 ME-TRAP and 2x10^8 pfu MVA ME-TRAP vaccines, 8 weeks apart, and then a CHMI intradermally (ID) by inoculation of 22,500 PfSPZ Challenge, 4 weeks later.
  Interventions: Biological: ChAd63/MVA ME-TRAP; Biological: intradermal injection (ID) or direct venous injection (DVI) of PfSPZ Challenge
- Group 3 (Experimental): Group 3 adults (n=14) will be receiving, 4 weeks apart, three doses of 10µg R21 /50µg Matrix M vaccine, and a CHMI intravenously (DVI) by inoculation of 3,200 PfSPZ Challenge.
  Interventions: Biological: R21/Matrix-M; Biological: intradermal injection (ID) or direct venous injection (DVI) of PfSPZ Challenge
- Group 4 (Experimental): Group 4 adults (n=18) will be the control group receiving no vaccine, only a CHMI intradermally (ID) by inoculation of 22,500 PfSPZ Challenge.
  Interventions: Biological: intradermal injection (ID) or direct venous injection (DVI) of PfSPZ Challenge

INTERVENTIONS:
Biological: R21/Matrix-M — R21: Protein particle malaria vaccine candidate in Matrix-M: Saponin based vaccine adjuvant.
  Arms: Group 1; Group 3
Biological: ChAd63/MVA ME-TRAP — ChAd63, chimpanzee adenovirus serotype 63; ME-TRAP, multiple epitope string fused to the thrombospondin-related adhesion protein; MVA, modified vaccinia Ankara.
  Arms: Group 2
Biological: intradermal injection (ID) or direct venous injection (DVI) of PfSPZ Challenge — PfSPZ Challenge: cryopreserved Plasmodium falciparum sporozoites.

SUMMARY:
This is a phase IIb clinical trial in malaria-exposed individuals to assess the immunogenicity, safety and efficacy of the two vaccines in the context of controlled human malaria infection, P. falciparum sporozoite challenge (PfSPZ Challenge).

DETAILED DESCRIPTION:
A total of 64 participants will be enrolled for challenge and divided into four groups as follows:

* 20 participants to receive R21/Matrix M (R21/MM) with intradermal PfSPZ Challenge;
* 20 participants to receive viral-vectored ME-TRAP with intradermal PfSPZ Challenge;
* 10 participants to receive R21/MM with direct venous inoculation PfSPZ Challenge; and
* 14 participants comprising of the control group with intradermal PfSPZ Challenge.

Blood tests and clinical assessments will be conducted to screen out participants with health conditions that may impact participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Non-pregnant, non-lactating adult female or adult male
* Agreement to refrain from blood donation during the study
* Use of effective method of contraception for the duration of study for female participants. For those with no contraception, they will be referred for contraception at the relevant health facility. For female participants, we will ask them to attend with their family planning records for verification. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined oral contraceptives; injectable progestogen; implants of etenogestrel or levonorgestrel; intrauterine device or intrauterine system; male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository); and male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository)
* Provide written informed consent
* Plan to remain resident in the study area for 1 year following first dose of vaccination

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the study clinicians
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Sickle cell disease
* Any history of anaphylaxis in relation to vaccination
* Clinically significant laboratory abnormality as judged by the study clinician
* Blood transfusion within one month of enrolment
* Haemoglobin less than 11.3 g/dl for men and less than 10g/dl for in women, where judged to be clinically significant in the opinion of the investigator.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG)
* Use of systemic antibiotics with known antimalarial activity within 30 days of administration of PfSPZ Challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Women only; pregnancy, or an intention to become pregnant a day before challenge i.e. at C-1
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* Confirmed parasite positive by PCR a day before challenge i.e. at C-1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited local and systemic reactogenicity signs and symptoms, and unsolicited adverse events | Solicited AEs are collected for 7 days post vaccination and unsolicited AEs for 28 days post vaccination
  Assessing the safety and reactogenicity of adjuvanted R21/MM and heterologous prime- boost regime of ChAd63-MVA ME-TRAP in healthy adult volunteers
Occurrence of P. falciparum parasitemia assessed by PCR, and parasite density dynamics assessed by PCR, against malaria sporozoite challenge | up to 3 months after malaria sporozoite challenge
  To assess the safety of intradermal sporozoite infection dose in semi-immune healthy adult volunteers
Occurrence of P. falciparum parasitemia, assessed by qPCR | from vaccination day up to 90 days after malaria sporozoite challenge
  To assess the efficacy of adjuvanted R21 and heterologous prime- boost regime of ChAd63-MVA ME-TRAP against malaria sporozoite challenge, in healthy adult volunteers

SECONDARY OUTCOMES:
To measure cellular immunogenicity assessed by ELISPOT | from vaccination day up to 90 days after malaria sporozoite challenge
  Assessing cellular immunogenicity by ELISPOT to enumerate IFN-ƴ producing T cells
To measure humoral immunogenicity assessed by ELISA | from vaccination day up to 90 days after malaria sporozoite challenge
  Assessing humoral immunogenicity by ELISA to quantify antibodies to the vaccine components CS, NANP, TRAP and HBsAb.
Parasite density dynamics assessed by qPCR | up to 3 months after malaria sporozoite challenge
  To assess any differences in efficacy estimates with ID versus DVI challenge in individuals receiving R21/MM

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI/Wellcome Trust Programme, Centre for Geographic Medicine Research - Coast, Kilifi, Kenya

REFERENCES:
- [Derived] Kapulu MC, Orenge F, Kimani D, Kibwana E, Kibet H, Mutahi M, Datoo MS, Bellamy D, Musembi J, Ngoto O, Rashid H, Akinyi S, Mwatasa MH, Nyamako L, Keter K, Gatheru R, Mutiso A, Musyoki J, Mwacharo J, Abebe Y, James ER, Billingsley PF, Ngetsa C, Mosobo M, Makale J, Tawa B, Wamae K, Ochola-Oyier LI, Lawrie A, Ramos-Lopez F, Roberts R, Richie TL, Sim BKL, Hoffman SL, Ewer KJ, Hill AVS, Hamaluba M, Bejon P. Malaria vaccine protection against intradermal or venous parasites: a randomized phase 2b human challenge trial. Nat Med. 2026 Jan;32(1):178-185. doi: 10.1038/s41591-025-04107-6. Epub 2026 Jan 6. PMID 41495411